CLINICAL TRIAL: NCT07141355
Title: Microcirculatory Effects of Empagliflozin in Patients With Cardiogenic Shock: an Ancillary Pilot Study of the EMPASHOCK Trial
Brief Title: Empagliflozin's Microcirculatory Effects in Cardiogenic Shock: an Ancillary Pilot Study of the EMPASHOCK Trial
Acronym: EMPAmicroSHOCK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 9357
Record Dates: First submitted 2025-08-04; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Cardiogenic Shock
Keywords: Cardiogenic Shock; Acute Heart failure; Heart failure
MeSH Terms: conditions — Shock, Cardiogenic; Heart Failure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient in cardiogenic shock under empagliflozin (Active Comparator): Subgroup of patients from the EMPASHOCK trial, in which microcirculation parameters will be evaluated at inclusion (before being under empagliflozin treatment) and again after 48 hours.
  Interventions: Diagnostic Test: microcirculation using the video microscopy tool.
- Patient in cardiogenic shock without empagliflozin (Sham Comparator): Subgroup of patients from the EMPASHOCK trial, without empagliflozin, in which microcirculation parameters will be evaluated at inclusion and again after 48 hours.
  Interventions: Diagnostic Test: microcirculation using the video microscopy tool.

INTERVENTIONS:
Diagnostic Test: microcirculation using the video microscopy tool. — The study intervention is the assessment of microcirculation using the video microscopy tool.
  This study's primary purpose is to perform this specific diagnostic procedure-measuring microcirculatory parameters with the CytoCam-IDF device-at two distinct time points: at inclusion (H0) and again 48 hours later (H48).
  The administration of empagliflozin (or not), which is pa and 48 hours after initiating empagliflozin treatment, microcirculatory data will be collected using a videomicroscope. A camera, roughly the size of a large pen, is placed under the patient's tongue for a few seconds to acquire images of the sublingual microcirculation. The entire image acquisition process takes less than 5 minutes and is unaffected by whether the patient is intubated.
  Images are then analyzed in real-time by the MicroTools software, which calculates key microcirculatory parameters.
  All anonymized images are stored on a dedicated, password-protected computer accessible only to the investigators.

SUMMARY:
Despite advancements in treatment, the mortality rate for cardiogenic shock (CS) remains high at around 50%. The EMPULSE-HF trial showed that early introduction of empagliflozin in stabilized patients with acute heart failure led to a composite benefit in mortality, rehospitalization, and quality of life.

Growing evidence suggests that cardiogenic shock isn't just a problem of systemic macrocirculation (blood pressure, cardiac output). It also involves significant abnormalities in the systemic microcirculation. In fact, these microcirculatory parameters have proven to be better predictors of patient outcomes than traditional macrocirculatory measures.

Given its known vasculo-protective effects on the endothelium, empagliflozin may have a beneficial impact on the microcirculation, potentially explaining its positive effects in cardiogenic shock.

This study will explore this hypothesis by analyzing the microcirculation in real-time using the CytoCam-IDF imaging videomicroscope and its MicroTools software. The goal is to gain a deeper understanding of how empagliflozin affects the microcirculation during cardiogenic shock.

DETAILED DESCRIPTION:
This ancillary pilot study, conducted in an ICU, investigates the real-time microcirculatory effects of empagliflozin in patients with cardiogenic shock (CS). The study aims to determine if the drug improves microcirculation, which is a known predictor of patient outcomes in CS.

Upon a patient's inclusion in the main EMPASHOCK trial, consent for this ancillary study is obtained from the patient's family, with direct patient consent sought later if their condition improves.

The study involves two data collection points:

Baseline (H0): Before empagliflozin administration, a videomicroscope is used to capture sublingual microcirculation images. These images are analyzed using MicroTools software to measure key microcirculatory parameters. Standard macrocirculatory parameters (blood pressure, cardiac output) are also recorded.

48 Hours (H48): The same microcirculatory and macrocirculatory data are collected again to assess changes following treatment.

For patients in the non-empagliflozin group, assessment will be perform at inclusion (H0) and at H48.

The study's primary outcomes are the changes in these parameters over 48 hours, along with the patient's survival status at day 28.

ELIGIBILITY:
Inclusion Criteria:

* Patient included in the main EMPASHOCK study
* Patient has signed a consent form for the ancillary study
* Patient is over 18 years old
* Hospitalized in the Intensive Care Unit for cardiogenic shock*
* Has been or is on catecholamines for at least 12 hours for the treatment of cardiogenic shock**
* Patient has the ability to take tablets orally
* Person is affiliated with or a beneficiary of a social security system

Exclusion Criteria:

* • GFR < 20 ml/min/1.73m²

  * Chronic dialysis
  * Patient on SGLT2 inhibitors prior to ICU admission
  * Known allergy to SGLT2 inhibitors or any of their excipients (in particular, patients with hereditary galactose intolerance, total lactase deficiency, or glucose-galactose malabsorption syndrome).
  * Patient on lithium
  * Patient with type 1 diabetes
  * Patient in shock due to another cause or moribund patient (IGS 2 > 90)
  * Cardiogenic shock cases excluded in the EMPASHOCK study: a. Heart transplant recipient or on a transplant list. b. Peripartum, adrenergic, valvular, restrictive, or post-embolic cardiomyopathy. c. Related to cardiotropic drug intoxication. d. Secondary to cardiac arrest where the patient remains comatose before inclusion.
  * Woman of childbearing age without effective contraception
  * Person referred to in Articles 10, 31, 32, 33, and 34 of EU Regulation 536/2014, specifically:
* Pregnant woman, woman in labor, or breastfeeding mother
* Minor person (not emancipated)
* Adult person subject to a legal protection measure (guardianship, curatorship, legal safeguard)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
The difference in the evolution of a parameter reflecting the microcirculation between the two groups at 48 hours post-randomization. | Comparison between Day 0 and 48 hours
  To estimate the effect of the early introduction of empagliflozin, in addition to usual care versus usual care alone, at 48 hours post-randomization, on sublingual microcirculation.(functional capillary density (FCD)) with the CytoCam-IDF imaging videomicroscope and its MicroTools software

SECONDARY OUTCOMES:
Correlation between microcirculation parameters and macrocirculation parameters. | Comparison between Day 0 and 48 hours
  Cardiac power index
The difference in the evolution of other microcirculation parameters between the two groups at 48 hours. | Comparison between Day 0 and 48 hours
  Total vessel density (TVD)
The difference in the evolution of other microcirculation parameters between the two groups at 48 hours. | Comparison between Day 0 and 48 hours
  Proportion of perfused vessels (PPV)
The difference in the evolution of other microcirculation parameters between the two groups at 48 hours. | Comparison between Day 0 and 48 hours
  Functional capillary density (FCD),
The difference in the evolution of other microcirculation parameters between the two groups at 48 hours. | Comparison between Day 0 and 48 hours
  Red blood cell mean velocity (RBCv)
The difference in the evolution of other microcirculation parameters between the two groups at 48 hours. | Comparison between Day 0 and 48 hours
  Per-capillary microcirculatory flow index (MFI)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France